CLINICAL TRIAL: NCT05393505
Title: Fast-track Absolute Neutrophil Count in Suspected Neutropenic Fever (The FRANCiS-NF Trial): A Single-centre, Pragmatic, Open-label, Randomised, Controlled Trial
Brief Title: Fast-track Blood Test for Suspected Fever by Deficiency of a Kind of White Blood Cells As Main Defense Against Infection
Acronym: FRANCiS-NF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC2178HKU1
Record Dates: First submitted 2021-12-22; First posted 2022-05-26 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Neutropenic Fever
Keywords: febrile neutropenia; emergency department; cancer; adult; sepsis; randomized controlled trial; antibiotic stewardship; clinical laboratory services; chemotherapy; hematopoietic stem cell transplantation
MeSH Terms: conditions — Febrile Neutropenia; Emergencies; Neoplasms; Sepsis | interventions — Meropenem; Levofloxacin; Amoxicillin-Potassium Clavulanate Combination; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: This is a single-center, pragmatic, open-labelled, randomized, controlled trial with 1:1 parallel-group assignment, which aims to establish superiority in antibiotic stewardship.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast-tRack Absolute Neutrophil Count (FRANC) Protocol (Experimental): Patient's blood sample will be expedited for complete blood count with differentials. Intravenous antibiotic is given depending on absolute neutrophil count. If neutropenia is present, broad-spectrum antibiotic (meropenem 1 g or levofloxacin 500 mg) will be given after septic workup within 1 hour of registration in emergency department before transfer to wards. If absent, antibiotic according to "Hospital Authority Interhospital Multi-disciplinary Programme on Antimicrobial ChemoTherapy (IMPACT)" with reference to previous bacterial sensitivity pattern, or amoxiclav 1.2 g if not specified, will be given. Other interventions are given according to clinical needs. The regimen is continued until clinicians recommend an alternative antimicrobial based on clinical grounds, or detection of other pathogens which indicate another antimicrobial.
  Interventions: Drug: Meropenem Injection; Drug: Levofloxacin; Drug: Amoxicillin Clavulanate; Drug: Antibiotic
- Standard of Care (Active Comparator): The control group refers to the existing clinical pathway which guides management of adult patients with suspected NF in ED. Without information of absolute neutrophil count, Meropenem 1 g IV bolus (or Levofloxacin 500 mg IV infusion over 1 hour if Penicillin-allergic) will be given within 1 hour of ED registration after septic workup. Other interventions are given according to clinical needs.
  Subsequent treatment in wards will be determined by doctor's clinical judgement, on a personalised basis. Each patient will be assessed by a parent team member. There is no standardised antibiotic de-escalation protocol in place, but it is a usual practice to continue Meropenem or Levofloxacin injections until clinical improvement, rising ANC, and negative culture results. After that it will be replaced with an antibiotic with a narrower spectrum, such as oral Amoxiclav, before discharge.
  Interventions: Drug: Meropenem Injection; Drug: Levofloxacin

INTERVENTIONS:
Drug: Meropenem Injection — Given if patient has no known allergies at 1 g IV bolus within 1 hour of ED registration, then every 8 hours
Drug: Levofloxacin — Given if patient is allergic to beta lactam at 500 g IV in 100 mL 0.9% sodium chloride solution, infused over 1 hour started within 1 hour of ED registration, then every 24 hours. If the patient can tolerate oral drugs, 500 mg daily after the first IV dose.
Drug: Amoxicillin Clavulanate — Given if patient has no known allergies at 1.2 g IV bolus within 1 hour of ED registration, then every 8 hours. If the patient can tolerate oral drugs, 1 g twice daily after the first IV bolus.
  Other Names: Augmentin
  Arms: Fast-tRack Absolute Neutrophil Count (FRANC) Protocol
Drug: Antibiotic — Any antibiotic for empirical therapy of common infections as recommended by the fifth version of "Hospital Authority Interhospital Multi-disciplinary Programme on Antimicrobial ChemoTherapy (IMPACT)" guideline, with reference to previous bacterial sensitivity pattern
  Other Names: IMPACT guideline
  Arms: Fast-tRack Absolute Neutrophil Count (FRANC) Protocol

SUMMARY:
This is a comparative study for adult participants with cancer who are suspected to have neutropenic fever (or fever with low neutrophil count) in emergency department. Neutrophil is a kind of defensive white blood cell combating against infection, especially by bacteria and fungi. Low neutrophil can be part of the disease progress or secondary to some cancer treatment. These participants are at high risk of developing infection-related complications including death.

Currently a dedicated clinical pathway has been in place in emergency department for suspected neutropenic fever, which offers fast-track medical consultation, blood tests and a very strong antibiotic (meropenem) as the first choice within 1 hour of registration. However, majority of such participants' neutrophil counts are not low. Most of them have no bacterial infection in the body, and have unremarkable short hospital stays. Early administration of meropenem in the majority of cases may be unnecessary and imposes risk of developing antibiotic resistance.

This study attempts to answer the question, "In adult participants with cancer presenting to emergency department with suspected neutropenic fever, when compared with conventional treatment, can a new protocol guided by fast-track neutrophil count reduces prescription of meropenem?" Agreed participants will be randomly assigned to the conventional treatment group, or the new treatment group. For those who are assigned to the new treatment group, blood will be taken and sent to the hospital laboratory for urgent analysis of neutrophil count. Participants with proven low neutrophil counts will still receive meropenem, while those without low neutrophil counts will receive less strong antibiotic according to their clinical diagnoses, such as Augmentin. They will be followed up on the first 7 days, and then on the 14th, 30th, 90th, and 180th days after recruitment. Comparisons will be made to see how much less meropenem will be prescribed, and whether more serious adverse events will happen. The study is expected to take 37 months to complete. Duration of data collection, including the day of last follow up, is estimated to be 33 months.

DETAILED DESCRIPTION:
1. Background

1.a. Burden of neutropenic fever Neutropenic fever (NF), or febrile neutropenia, is characterised by high body temperature and low absolute neutrophil count (ANC) following myelosuppressive cancer treatment.[1] It occurs in 5 - 10 percent of patients with early-stage solid tumours, 20 - 25 percent with non-leukaemic haematological cancers, 85 - 95 percent with acute leukaemia,[2] and 13 - 21 percent with metastatic solid tumours.[1] It is more common after the first cycle of chemotherapy. 7.83 per 1,000 cancer patients were hospitalised for NF annually in the United States (US).[3] With earlier cancer recognition, and more prescriptions of chemotherapeutic agents and targeted therapies, the figures are expected to rise.

NF is associated with unplanned chemotherapy interruptions and relative dose intensity (RDI) reductions more than 15 percent, which undermine treatment success rates and overall survival.[2] When complicated by neutropenic sepsis, a dysregulated host response against infection, NF becomes an oncological emergency. The mortality rate is 3 - 18 percent following complications e.g. hypotension, respiratory failure, encephalopathy, cardiac failure and arrhythmia, renal failure, haemorrhage, and admission to intensive care unit (ICU).[4] Risk factors of life-threatening infections are severe neutropenia, protracted neutropenia, and splenectomy.[5] Mortality risk increases with advanced age, comorbidities, clinically documented infection, bacteraemia, leukaemia and lung cancer as underlying malignancies.[4,6]

The cost of managing NF remains substantial for healthcare systems worldwide. The mean direct hospitalisation costs in the US, Germany, and Singapore were US$19,110 (1995-2000), €3,950 (2005-2006), and US$4,913 (2009-2012) respectively.[6-8] Higher costs are associated with inpatient treatment, comorbidities, discharge, deaths, male sex, and infection.[9]

1.b. Diagnostic criteria NF is defined by 1) single oral temperature ≥ 38.3 degree Celsius (101ºF), or ≥ 38.0 degree Celsius (100.4ºF) sustained over 1 hour; and 2) ANC < 1.0 x 109/L ("moderate" neutropenia). Neutropenia becomes "severe", "profound" and "protracted" if ANC < 0.5 x 109/L, < 0.1 x 109/L, and lasts for more than one week, respectively.[10] This definition applies to oncological and haematological participants only.

1. c. Aetiology Neutrophils are recruited early during the acute phase of bacterial and fungal infections.[11] Fever may be the only manifestation of infection during neutropenia because the typical signs of inflammation are obscured. Neutropenia is usually acquired by myelosuppressive cancer treatments, and pre-engraftment phases of haematopoietic stem cell transplantation (HSCT). Bone marrow failure and defective neutrophil maturation are other possible mechanisms.[12]

   NF can have infectious and non-infectious causes. Fever of unknown origin, chemotherapy-related oral mucositis, tumour-related cytokine release, transfusion-related reaction, drug reaction, graft-versus-host disease, and thromboembolism are common non-infective causes.[13] 30 - 50 percent are infections by clinical presentation or microbiology,[14] whilst only 20 - 30 percent are microbiologically documented infections.[15] Bloodstream infections, bacterial translocation from respiratory tract and perianal region, and central venous catheter are major sources.

1.d. Situation in Hong Kong Local public emergency departments (EDs) have implemented clinical pathways for suspected NF, which expedite medical consultation, septic workup, and broad-spectrum antibiotics such as Meropenem or Piperacillin/Tazobactam. The target time from ED registration to antibiotic administration, or Door-To-Antibiotic (DTA) time, is within 1 hour disregarding ANC, in line with international guidelines.[16-18] DTA times are shortened after implementing clinical pathways in local ED.[19] Local epidemiology, antibiotic sensitivity patterns, and healthcare cost in managing NF are understudied. It has been shown that inadequate antibiotic regimen was more significantly associated with ICU admissions and mortality than longer DTA times. Presence of sepsis or septic shock, prior colonisation with drug resistant strains, and risk stratifying indices, are criteria to judge antibiotic adequacy.[20]

1. e. Antibiotic stewardship for cancer participants Participants with cancer are frequently exposed to antibiotics for treatment and prophylaxis, therefore they are more vulnerable to multi-drug resistance, and are in special need for antibiotic stewardship.[21] Broad-spectrum antibiotics are often started empirically in ED for suspected NF, assuming infection by drug-resistant bacteria. However, clinicians may not proactively de-escalate subsequent antibiotics. Prolonged exposures to parenteral broad-spectrum antibiotic impose risks of nosocomial infection and injection site complications.

   Gram-negative bacilli are more frequent in neutropenia. Staphylococcus aureus, Acinetobacter and Enterobacter species are more frequent in non-neutropenic bloodstream infections.[22] More drug resistant (MDR) strains, such as Extended-spectrum Beta-lactamase (ESBL)-producing Enterobacteriaceae, MDR Pseudomonas aeruginosa, and MDR Acinetobacter were isolated from neutropenic patients in a survey in China.[23]
2. Research (PICO) question In adult participants with cancer presenting to the ED with suspected NF, can an ED protocol guided by Fast-tRack Absolute Neutrophil Count (FRANC protocol) compared with conventional care guided by clinical suspicion alone improve safe antibiotic stewardship?
3. Objective and purpose

3.a. Objectives

In adult participants presenting to the ED with suspected NF:

* To investigate the effectiveness of the FRANC protocol to improve antibiotic stewardship by restricting meropenem use except for confirmed neutropenic or clinically unstable participants; and
* To investigate the safety of the FRANC protocol. 3.b. Primary hypothesis In participants presenting to ED with suspected NF, the FRANC protocol significantly reduces unnecessary use of Meropenem compared with normal Standard of Care (SoC).

  3.c. Secondary hypothesis In participants presenting to ED with suspected NF, there is no significant difference between those receiving the FRANC protocol and those receiving SoC for serious adverse events including death.

  4. Methods

  4.a. Participants 4.a.1. Target population This trial targets to adult participants attending ED because of fever, who are at risk of neutropenia related to cancer therapies and underlying conditions.

  4.a.2. Study location The trial will be conducted in the ED of Queen Mary Hospital with an average annual attendance of 125,000. The hospital is a tertiary referral centre for HSCT and oncological services which received more than 500 adults with suspected NF via the ED in 2019.

  4.a.3. Recruitment and screening Alert cards are routinely issued to participants at risk of neutropenia during follow-ups in Clinical Oncology and Haematology centres. They are reminded to visit EDs as soon as possible when fever occurs. A neutropenic risk alert is set to pop up in the Clinical Management System (CMS) that is shared among all public medical facilities. It is valid for 6 weeks from the last chemotherapy against solid tumours, or lifelong for haematological malignancies, and HSCT.

When febrile participants with valid alerts attend, the triage nurse will declare "1 - Critical" or "2 - Emergency" categories according to clinical state. Consultations by emergency physician will start within 15 minutes. Participants who receive cancer treatment in other medical facilities will also be included if they meet the same criteria.

Participants will then be screened for eligibility by trained research staff for inclusion and exclusion criteria in the ED. Potential participants will be invited to provide informed consent in written, signed, and dated forms. They can decline at any time.

4.a.4. Sample size For antibiotic stewardship A sample size of 344 participants (172 per group) will achieve 80 percent power to detect a superiority difference between two group rates of meropenem prescription. We set the superiority margin at 10 percent and assume that the control group has Meropenem usage rate of 91.8 percent (based on preliminary data) and 71.8 percent for intervention group. The calculation is based on a one-sided Z test at the significance level of 0.05.

4.a.5. Randomisation & allocation concealment We aim to achieve balanced treatment assignments in 1:1 ratio with simple randomisation by a computer-generated code list. The code is not broken until the last participant is enrolled and has completed 180 days of follow-up. It will be implemented using independent electronic case data files to ensure allocation concealment.

4.b. Data processing and analysis 4.b.1. Data processing All data will be entered electronically by research staff to password-protected, secured, web-based system with tailor-made recording forms using tablet computers. 5 percent of all data will be checked for accuracy. All hard copies will be restricted and locked in unit cabinets. All prevailing regulations by The University of Hong Kong and the Hospital Authority will be strictly followed. An audit trail will be made to include the number of participants screened, approached, recruited, and excluded (with reasons). Participant and clinical staff responses, and data completeness will be evaluated.

4.b.2. Data analysis 4.b.2.a. Primary analysis Baseline characteristics between two groups will be assessed for potential imbalances, which will be adjusted for when comparing outcomes. Intention-to-treat (ITT) analysis will be used by imputing all non-responses at follow-up with baseline values, which yields more conservative estimates of effect sizes. The missing data for the primary outcome is expected to be < 1 percent because most data is retrievable from electronic participant records with electronic time stamps. Statistical analysis will be done using Statistical Package of Social Sciences (SPSS) version 26 (IBM SPSS Statistics, New York, US) with biostatistician support.

Main effect: Intervention vs. Control on proportion of participants receiving Meropenem in 7 days using Chi-squared test.

4.b.2.b. Secondary analyses

* All secondary outcomes at different time points using generalised mixed effect model for multiple intra-participant and inter-participant observations. Main and interaction effects will be assessed.
* Subgroup analysis to primary outcome based on age, gender, type of cancer/ conditions, disease status, therapy received, time interval from last chemotherapy or HSCT to ED registration, at 30, 60, 90 days (4) Sensitivity of ITT and per-protocol analyses for pre-defined co-variates, missing data (including participants lost to follow-up), will be done. Imputation method will depend on actual pattern of missing data.
* If the attrition rate is more than 5 percent, risks of attribution bias and influence to statistical power will be assessed.
* Complication rates over time will be compared with Poisson mixed effects models. Uses of inotrope, mechanical ventilation, renal replacement therapy, and ICU are analysed against mortality using appropriate survival analyses with time to event data.

ELIGIBILITY:
Inclusion Criteria:

* Age criteria: 18 years old or above; AND
* Body temperature criteria: Tympanic temperature ≥ 38.3 degree Celsius (100.9 degree Fahrenheit) within 24 hours before emergency department registration; AND
* Chemotherapy timeframe criteria: Last chemotherapy or targeted therapy within 6 weeks for any solid tumor, or in any period following therapies against leukemia, lymphoma, myelodysplastic syndrome, aplastic anemia, multiple myeloma, or recipient of hematopoietic stem cell transplantation; AND
* Modified Early Warning Score (MEWS) ≤ 4

Exclusion Criteria:

* Unable to provide informed consent
* Previous enrolment to this trial within 180 days, or without current resolution of the first episode
* Enrolment to other interventional trials within 187 days
* Sepsis or septic shock
* Suspected central nervous system infection
* Severe desaturation (SpO2 < 88% in room air for patients with chronic obstructive pulmonary disease, severe chest wall or spinal disease, neuromuscular disease, severe obesity, cystic fibrosis, bronchiectasis; or < 94% in room air without)
* Currently on prophylactic antibiotic
* Any antibiotic treatment for > 48 h within 1 week
* Known human immunodeficiency virus infection
* Primary humoral immunodeficiency
* Complement deficiency
* Asplenia
* Vulnerable subjects (illiterate, pregnancy, mentally incapacitated, impoverished, prisoner, subordinate or students of investigators, ethnic minorities)
* Research staff not available
* Unable to randomize within 1 hour of emergency department registration
* Inter-hospital transfer
* Scheduled "clinical" admissions
* Body temperature not documented
* Blood sample not taken in emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Antibiotic stewardship as assessed by proportion of participants receiving Meropenem | Up to 7 days post-randomisation
  Proportion of participants in each group receiving Meropenem

SECONDARY OUTCOMES:
Clinically and/or microbiologically documented infections | Up to 15 days post-randomisation
  Rate and type of documented infective focus
Time to clinical improvement | Up to 15 days post-randomisation
  * Days to defervescence (body temperature less than 38 degree Celsius)
  * Days to resolution of symptoms and signs of infection
Incidence of adverse events requiring emergency interventions | Up to 15 days post-randomisation
  * Hypotension (systolic blood pressure < 90 mmHg)
  * Respiratory failure (partial pressure of oxygen in arterial blood < 60 mmHg, or 8 kilopascal, adjusted for hyperventilation)
  * Altered mental state (Glasgow Coma Scale < 15)
  * Congestive heart failure documented radiologically
  * Acute kidney injury (serum creatinine > 2x baseline, or estimated glomerular filtration rate (eGFR) > 50 percent increase from baseline, or urine output < 0.5 mL/kg/h x 12 h)
  * Acute liver failure (International Normalised Ratio (INR) > 1.5 in non-warfarin user, hepatic encephalopathy, total bilirubin > 85.5 µmol/L or 5 mg/dL)
  * Rate of therapeutic failure (recurrence of fever after defervescence)
Rate of life-saving interventions | Up to 15 days post-randomisation
  * Rate of inotrope/ vasopressor use
  * Rate of assisted / mechanical ventilation
  * Rate of renal replacement therapy
  * Rate of 3 or more units of blood transfusion for haemorrhage
  * Rate of additional antimicrobial treatment
  * Rate of Intensive Care Unit (ICU) admission
Length of hospital stay | Up to 180 days post-randomisation
  Total in-hospital days from the time of index ED admission
Proportion of participants with changes in chemotherapy schedule | Up to 180 days post-randomisation
  Changes in chemotherapy schedule following index admission (postponement, dose reductions, participant defaults)
Unplanned readmission rate | Up to 30 days post-randomisation
  Rates of any readmission except for planned chemotherapy
Overall survival | Up to 180 days post-randomisation
  Time from the day of randomisation to the date of death, all-cause or infection-related
Antibiotics administered | Up to 180 days post-randomisation
  Type and route of antibiotics administered, from the time of randomisation to hospital discharge, or from the time of randomisation to the expected date of completion of prescribed antibiotic courses after discharge, whichever the later
Mean total dose of antibiotics used | Up to 180 days post-randomisation
  Mean total dose of antibiotics used, in milligrams, from the time of randomisation to hospital discharge, or from the time of randomisation to the expected date of completion of prescribed antibiotic courses after discharge, whichever the later
Hospital antibiotics use as total days of antibiotic therapy (DOT) | Up to 180 days post-randomisation
  Total days of therapy (DOT) per admission - the unit measure is defined as one day in which a patient is given a drug, regardless of dose per admission.
Hospital antibiotics use as defined daily dose (DDD) per admission | Up to 180 days post-randomisation
  Defined daily dose (DDD) per admission is the assumed average maintenance dose, in milligrams, per day for a drug used for its main indication.
Microbiological safety as assessed by development of antibiotic resistance | Up to 180 days post-randomisation
  Development of resistance, defined as clinical isolates resistant to antibiotics previously used in the febrile episode. Surveillance sampling will not be conducted.
Health related quality of life as assessed by Functional Assessment of Cancer Therapy - General (FACT-G) | Up to 180 days post-randomisation
  Physical, social, emotional and function well being of participants will be evaluated using the standardised 27-item questionnaire, "Functional Assessment of Cancer Therapy - General" (FACT-G).
Health related quality of life as assessed by Functional Assessment of Cancer Therapy - Neutropenia (FACT-N) | Up to 180 days post-randomisation
  Physical, social, emotional and function well being of participants will be evaluated using the Functional Assessment of Cancer Therapy - Neutropenia (FACT-N). It is a modified version of the Functional Assessment of Cancer Therapy - General (FACT-G) with the Neutropenia subscale, which is targeted for adult cancer patients with neutropenia.
Financial Toxicity related to cancer and its treatment as assessed by Functional Assessment of Chronic Illness Therapy - COprehensive Score for financial Toxicity (FACIT-COST) | Up to 180 days post-randomisation
  Financial toxicity is evaluated using the Functional Assessment of Chronic Illness Therapy - COprehensive Score for financial Toxicity (FACIT-COST). The COST is a patient-reported outcome measure that describes the financial distress experienced by cancer patients. The FACIT System screens for financial toxicity and to provide a global summary item for financial toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Hudson Rainer, MBBCh; MRCP, Principal Investigator — Department of Emergency Medicine, Li Ka Shing Faculty of Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weycker D, Li X, Edelsberg J, Barron R, Kartashov A, Xu H, Lyman GH. Risk and Consequences of Chemotherapy-Induced Febrile Neutropenia in Patients With Metastatic Solid Tumors. J Oncol Pract. 2015 Jan;11(1):47-54. doi: 10.1200/JOP.2014.001492. Epub 2014 Dec 9. PMID 25491042
- [Background] Culakova E, Thota R, Poniewierski MS, Kuderer NM, Wogu AF, Dale DC, Crawford J, Lyman GH. Patterns of chemotherapy-associated toxicity and supportive care in US oncology practice: a nationwide prospective cohort study. Cancer Med. 2014 Apr;3(2):434-44. doi: 10.1002/cam4.200. Epub 2014 Feb 17. PMID 24706592
- [Background] Caggiano V, Weiss RV, Rickert TS, Linde-Zwirble WT. Incidence, cost, and mortality of neutropenia hospitalization associated with chemotherapy. Cancer. 2005 May 1;103(9):1916-24. doi: 10.1002/cncr.20983. PMID 15751024
- [Background] Klastersky J, Ameye L, Maertens J, Georgala A, Muanza F, Aoun M, Ferrant A, Rapoport B, Rolston K, Paesmans M. Bacteraemia in febrile neutropenic cancer patients. Int J Antimicrob Agents. 2007 Nov;30 Suppl 1:S51-9. doi: 10.1016/j.ijantimicag.2007.06.012. Epub 2007 Aug 8. PMID 17689933
- [Background] Bodey GP, Buckley M, Sathe YS, Freireich EJ. Quantitative relationships between circulating leukocytes and infection in patients with acute leukemia. Ann Intern Med. 1966 Feb;64(2):328-40. doi: 10.7326/0003-4819-64-2-328. No abstract available. PMID 5216294
- [Background] Kuderer NM, Dale DC, Crawford J, Cosler LE, Lyman GH. Mortality, morbidity, and cost associated with febrile neutropenia in adult cancer patients. Cancer. 2006 May 15;106(10):2258-66. doi: 10.1002/cncr.21847. PMID 16575919
- [Background] Ihbe-Heffinger A, Paessens BJ, von Schilling C, Shlaen M, Gottschalk N, Berger K, Bernard R, Kiechle M, Peschel C, Jacobs VR. Management of febrile neutropenia--a German prospective hospital cost analysis in lymphoproliferative disorders, non-small cell lung cancer, and primary breast cancer. Onkologie. 2011;34(5):241-6. doi: 10.1159/000327711. Epub 2011 Apr 26. PMID 21577029
- [Background] Wang XJ, Wong M, Hsu LY, Chan A. Costs associated with febrile neutropenia in solid tumor and lymphoma patients - an observational study in Singapore. BMC Health Serv Res. 2014 Sep 24;14:434. doi: 10.1186/1472-6963-14-434. PMID 25252614
- [Background] Wang XJ, Lopez SE, Chan A. Economic burden of chemotherapy-induced febrile neutropenia in patients with lymphoma: a systematic review. Crit Rev Oncol Hematol. 2015 May;94(2):201-12. doi: 10.1016/j.critrevonc.2014.12.011. Epub 2014 Dec 31. PMID 25600838
- [Background] Taplitz RA, Kennedy EB, Bow EJ, Crews J, Gleason C, Hawley DK, Langston AA, Nastoupil LJ, Rajotte M, Rolston KV, Strasfeld L, Flowers CR. Antimicrobial Prophylaxis for Adult Patients With Cancer-Related Immunosuppression: ASCO and IDSA Clinical Practice Guideline Update. J Clin Oncol. 2018 Oct 20;36(30):3043-3054. doi: 10.1200/JCO.18.00374. Epub 2018 Sep 4. PMID 30179565
- [Background] Kobayashi SD, Voyich JM, Burlak C, DeLeo FR. Neutrophils in the innate immune response. Arch Immunol Ther Exp (Warsz). 2005 Nov-Dec;53(6):505-17. PMID 16407783
- [Background] Boxer L, Dale DC. Neutropenia: causes and consequences. Semin Hematol. 2002 Apr;39(2):75-81. doi: 10.1053/shem.2002.31911. PMID 11957188
- [Background] Pasikhova Y, Ludlow S, Baluch A. Fever in Patients With Cancer. Cancer Control. 2017 Apr;24(2):193-197. doi: 10.1177/107327481702400212. PMID 28441374
- [Background] Castagnola E, Mikulska M, Viscoli C. Prophylaxis and Empirical Therapy of Infection in Cancer Patients. Mandell, Douglas, and Bennett's Principles and Practice of Infectious Diseases. 2015:3395-3413.e2. doi: 10.1016/B978-1-4557-4801-3.00310-6. Epub 2014 Oct 31. PMCID: PMC7173426.
- [Background] Pizzo PA, Robichaud KJ, Wesley R, Commers JR. Fever in the pediatric and young adult patient with cancer. A prospective study of 1001 episodes. Medicine (Baltimore). 1982 May;61(3):153-65. doi: 10.1097/00005792-198205000-00003. No abstract available. PMID 7078399
- [Background] Taplitz RA, Kennedy EB, Bow EJ, Crews J, Gleason C, Hawley DK, Langston AA, Nastoupil LJ, Rajotte M, Rolston K, Strasfeld L, Flowers CR. Outpatient Management of Fever and Neutropenia in Adults Treated for Malignancy: American Society of Clinical Oncology and Infectious Diseases Society of America Clinical Practice Guideline Update. J Clin Oncol. 2018 May 10;36(14):1443-1453. doi: 10.1200/JCO.2017.77.6211. Epub 2018 Feb 20. PMID 29461916
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Background] Ko HF, Tsui SS, Tse JW, Kwong WY, Chan OY, Wong GC. Improving the emergency department management of post-chemotherapy sepsis in haematological malignancy patients. Hong Kong Med J. 2015 Feb;21(1):10-5. doi: 10.12809/hkmj144280. Epub 2014 Oct 10. PMID 25306894
- [Background] Peyrony O, Gerlier C, Barla I, Ellouze S, Legay L, Azoulay E, Chevret S, Fontaine JP. Antibiotic prescribing and outcomes in cancer patients with febrile neutropenia in the emergency department. PLoS One. 2020 Feb 28;15(2):e0229828. doi: 10.1371/journal.pone.0229828. eCollection 2020. PMID 32109264
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Velasco E, Byington R, Martins CA, Schirmer M, Dias LM, Goncalves VM. Comparative study of clinical characteristics of neutropenic and non-neutropenic adult cancer patients with bloodstream infections. Eur J Clin Microbiol Infect Dis. 2006 Jan;25(1):1-7. doi: 10.1007/s10096-005-0077-8. PMID 16424972
- [Background] Zhu J, Zhou K, Jiang Y, Liu H, Bai H, Jiang J, Gao Y, Cai Q, Tong Y, Song X, Wang C, Wan L. Bacterial Pathogens Differed Between Neutropenic and Non-neutropenic Patients in the Same Hematological Ward: An 8-Year Survey. Clin Infect Dis. 2018 Nov 13;67(suppl_2):S174-S178. doi: 10.1093/cid/ciy643. PMID 30423039
- [Background] So SN, Ong CW, Wong LY, Chung JY, Graham CA. Is the Modified Early Warning Score able to enhance clinical observation to detect deteriorating patients earlier in an Accident & Emergency Department? Australas Emerg Nurs J. 2015 Feb;18(1):24-32. doi: 10.1016/j.aenj.2014.12.001. Epub 2015 Jan 15. PMID 25601429
- See also: National Institute for Health and Care Excellence: Guidance. Neutropenic Sepsis: Prevention and Management of Neutropenic Sepsis in Cancer Patients — https://www.nice.org.uk/guidance/cg151
- See also: Reducing bacterial resistance with IMPACT - Interhospital Multi-disciplinary Programme on. Antimicrobial ChemoTherapy (version 5.0) — https://www.chp.gov.hk/files/pdf/reducing_bacterial_resistance_with_impact.pdf